CLINICAL TRIAL: NCT07019454
Title: Baystate Health Physician Sponsored - Investigational Device Exception: Physician Modified Endovascular Grafts for the Treatment of Elective, Symptomatic or Ruptured Juxtarenal Aortic Aneurysms
Brief Title: Physician Modified Endovascular Grafts for the Treatment of Elective, Symptomatic or Ruptured Juxtarenal Aortic Aneurysms
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baystate Medical Center (Other)
Responsible Party: Principal Investigator, Hazel Marecki, MD, Vascular Surgeon, Baystate Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2303212-3; G240287 (Other: FDA)
Record Dates: First submitted 2025-06-03; First posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Technical Sucess; Freedom From Type I and III Endoleaks at 12 Months; Freedom From Stent Graft Migration at 12 Months; Freedom From Aortic Aneurysm Enlargement at 12 Months; Freedom From Aortic Aneurysm Rupture or Conversion to Open Repair at 12 Months
Keywords: complex endovascular aortic aneurysm repair; PMEG; juxtarenal

STUDY DESIGN:
Intervention Model Description: Selected patients based on anatomic criteria will be offered to be included in the study and undergo repair with physician modified endografting only if they are deemed not to be a candidate for an alternative FDA approved endovascular aortic repair device.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Physician Modified Endograft Group (Experimental): Patients in this arm will undergo physician modified endovascular grafting of their juxtarenal aortic aneurysm
  Interventions: Device: Physician Modified Endografting

INTERVENTIONS:
Device: Physician Modified Endografting — This is the only intervention in the study
  Other Names: PMEG

SUMMARY:
Patients who are found to have an aneurysm (bulge) in the abdominal aorta, which is the blood vessel in your abdomen (belly) that supplies blood to most of your lower body, including major organs and your legs. As an aneurysm expands, the walls of the aorta become weak and may rupture (break open), causing a major loss of blood with a high risk of serious problems and death. To avoid this risk, doctors repair aneurysms by either open surgery (incision) or endovascular surgery (covered stents to channel the blood flow). Juxtarenal aneurysms (those that come close to the kidney arteries) present a unique challenge as they are more dangerous to repair by open therapy and do not fit the standard approved endovascular devices. The purpose of this study is to assess the effects of the physician-modified endovascular graft (PMEG) by collecting information about the performance of this investigational medical device.

The main graft looks like a pair of pants with very short legs. The top of the pants is placed in the aorta. Then, two smaller grafts go from the main graft and to your iliac arteries (the main arteries supplying blood to your abdomen and legs) to form the legs of the pair of pants. Each graft is packed into a small catheter (a long, flexible plastic tube) that is placed into your aorta through the femoral artery in your groin (top of your leg). The grafts are then placed in the correct position in your aorta by releasing them from the catheters. These grafts are investigational because the research physician has changed them to match patient anatomy (body make up) while protecting blood flow to important vessels. Once the grafts are attached inside the aorta, they will support the area of the aorta that is weakened and bulging.

Modifications of the graft will include between one and four holes (fenestrations) near the top of the graft. The holes allow the graft to be located above the renal arteries (the blood vessels that supply blood to your kidneys) without blocking the blood flow to them. One or more of the arteries will also be treated with a stent (metal wire tube) to help keep the arteries open and to keep the arteries connected to the holes that are made for the graft.

The device is custom modified for patient specific anatomy. The information collected from this study will be used to show how well patients do when treated with the modified graft, both immediately after surgery and over a long period of time. After the procedure, labs, CT imaging with contrast, XRays and ultrasounds will be done to check the graft at intervals 1 month, 6 months, 12 months and yearly for 5 years. These are standard surveillance studies performed on any endovascular aneurysm repair.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is ≥ 18 years of age
2. Patients who are male or non-pregnant female (females of child bearing potential must have a negative pregnancy test prior to enrollment into the study)
3. Patient or Legally Authorized Representative has signed an Institutional Review Board (IRB) approved Informed Consent Form
4. Patient has a juxtarenal abdominal aortic aneurysm that meets at least one of the following:

   1. An aneurysm with a maximum diameter of ≥ 5.5 cm for male (≥ 5.0 cm for female) or 2 times the normal diameter just proximal to the aneurysm using orthogonal (i.e., perpendicular to the centerline) measurements
   2. Aneurysm with a history of growth > 0.5 cm in 6 months
   3. Saccular aneurysm deemed at significant risk for rupture
   4. Symptomatic aneurysm
   5. Ruptured aneurysm
5. Patient has patent iliac or femoral arteries, with or without the use of conduit, that will allow endovascular access with the physician modified endovascular graft.
6. Patient has a suitable non-aneurysmal proximal aortic neck of ≥ 2 mm inferior to the most distal renal artery ostium.
7. Patient has a suitable non-aneurysmal distal iliac artery length (seal zone) of ≥ 15mm. The resultant repair should preserve patency in at least one hypogastric artery.
8. Patient has a suitable non-aneurysmal proximal aortic neck diameter between 20 and 32 mm, averaged across the diameters at the Celiac, SMA, at the lowest patent renal artery and at the midpoint of the renal arteries.
9. Patient has suitable non-aneurysmal distal common iliac diameters between 8 and 20 mm.
10. Patient has juxtarenal aortic neck angulation ≤ 60°
11. Target branch vessel diameter ≥ 5 mm.
12. Patient must be willing to comply with all required follow-up exams.

Exclusion Criteria:

1. Patient has a mycotic aneurysm or has an active systemic or local infection that may increase the risk of endovascular infection
2. Patient has unstable angina (defined as angina with a progressive increase in symptoms, new onset at rest or nocturnal angina, or onset of prolonged angina)
3. Patient has a major surgical or interventional procedure, not related to the endovascular repair, planned within +/- 30 days of the AAA repair.
4. Patient has history of an aortopathic connective tissue disease (e.g. Marfan's or Ehler's- Danlos syndrome).
5. Patient has a known hypersensitivity or contraindication to anticoagulation or contrast media that is not amenable to pre-treatment.
6. Patient has known allergy or intolerance to stainless steel, nitiol, or gold (gold-plated tungsten)
7. Patient has a body habitus that would inhibit X-ray visualization of the aorta
8. Patient has a limited life expectancy of less than 1 year
9. Patient is currently participating in another investigational device or drug clinical trial
10. Patient has other medical, social or psychological conditions that, in the opinion of the investigator, preclude them from receiving the pre-treatment, required treatment, and post- treatment procedures and evaluations.
11. Thrombus or excessive calcification within the neck of the aneurysm
12. Branch vessel stenosis ≥ 80 %
13. Patients treatable on label with FDA approved EVAR or FEVAR device and can wait for device availability.
14. Subject is willing and eligible to enroll in a manufacturer-sponsored study at the investigational site, or the subject is willing and eligible to participate in a study with a manufacturer-made device at another institution.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-06-03 (Actual); Primary Completion 2030-06-03 (Estimated); Study Completion 2035-06-03 (Estimated)

PRIMARY OUTCOMES:
Technical success | Periprocedural
  The physician was able to insert the delivery catheter and deliver the physician modified endovascular graft to the treatment site and preserve blood flow into the vessels intended to have blood flow preserved.
Freedom from Type I and III Endoleaks at 12 months | 12 months post-procedure
  Yes/No Type I or Type III Endoleak visualized on 12 month CT Angiography
Freedom from stent graft migration at 12 months | 12 months
  Yes/No stent migration at 12 months
Freedom from aortic aneurysm enlargement at 12 months | 12 months
  Yes/No Freedom from enlargement maximal aortic diameter
Freedom from aortic aneurysm rupture and conversion to open repair through 12 months | 12 months
  Yes/No freedom from

SECONDARY OUTCOMES:
Mortality | 30 days, 6 months, 12 months, and annually through 5 years
  Yes/No
Aneurysm related mortality | 30 days, 6 months, 12 months, and annually through 5 years
  Yes/ No
Aneurysm Rupture | 30 days, 6 months, 12 months, and annually through 5 years
  Yes/ No
Major Adverse Events | 30 days, 6 months, 12 months, and annually through 5 years
Renal failure with or without permanent dialysis | 30 days, 6 months, 12 months, and annually through 5 years
  Yes/No, with or without dialysis
Graft Infection | 30 days, 6 months, 12 months, and annually through 5 years
  Yes/ No

CONTACTS AND LOCATIONS:
Overall Officials: Hazel Marecki, MD, Principal Investigator — Baystate Medical Center
Locations (1):
- Baystate Medical Center, Springfield, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided
Unidentified data may be analyzed retrospectively with other hospitals who are conducting this study for data analysis and publication of results.